CLINICAL TRIAL: NCT06403033
Title: Evaluation of the Skeletal and Dentoalveolar Effects of Mini-implant-supported Twin-Block in Treating Growing Patients With Class II Division 1 Malocclusion: A Two-arm Randomized Controlled Clinical Trial
Brief Title: Mini-implant-supported Twin-Block in Treating Patients With Class II Division 1 Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-3-2024
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Orthodontic Appliance Complication; Malocclusion, Angle Class II, Division 1
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini-implant-supported Twin-Block (Experimental): Treatment will be done using the Mini-implant-supported Twin-block appliance until the correction is achieved.
  Interventions: Device: Mini-implant-supported Twin-Block
- Conventional Twin-Block group (Active Comparator): Treatment will be done using the Twin-block appliance until the correction is achieved.
  Interventions: Device: Twin-Block

INTERVENTIONS:
Device: Mini-implant-supported Twin-Block — Mini-implants will support the Twin-Block appliance during the functional treatment.
  Arms: Mini-implant-supported Twin-Block
Device: Twin-Block — This is the main appliance that will be used to correct the Class II deformity.
  Arms: Conventional Twin-Block group

SUMMARY:
Correcting the skeletal class II using functional appliances, whether removable or fixed, always leads to skeletal and alveolar effects. However, some of these effects are unfavorable, the most significant being the loss of support in the lower dental arch. This loss of support leads to an uncontrolled labial inclination of the lower incisors and mesial movement of the lower; these dentoalveolar effects impact the degree of skeletal correction that can be achieved. Therefore, this study aimed to evaluate the skeletal and dentoalveolar effects following the use of a mini-implant-supported Twin-Block appliance compared to the conventional Twin-Block.

DETAILED DESCRIPTION:
Many attempts have been made to modify the Twin-Block appliance to decrease the dentoalveolar effects, such as omitting the upper labial bow, including torquing spurs on the upper incisors, and adding acrylic capping on the lower incisors. However, these modifications have not been successful in eliminating the dentoalveolar effects. This is because the Twin-Block and other functional appliances are supported by teeth rather than bone. As a result, the components of the appliance exert force on the teeth while the mandible attempts to return to its natural resting position. No previous clinical trial described the use of the Twin-Block appliance supported by orthodontic mini-implants and the potential benefits of using mini-implants with Twin-Block in functional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The wrist radiograph (stage 4 S and stage 5 MP3 cap)
2. Skeletal Class II division 1 malocclusion caused by mandibular retrusion
3. ANB (5°- 9°)
4. SNB (72°- 77°)
5. overjet (5 - 8 mm),
6. Minimal crowding in dental arches (≤ 3 mm),
7. MM≤30°
8. lower second molars erupting.

Exclusion Criteria:

1. Previous orthodontic procedures.
2. Systemic diseases.
3. Temporal Mandibular Joint disorders.
4. Poor oral hygiene

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Change in the overjet | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from the upper central incisor edge to the labial surface of the lower central incisor (in mm).
Change in the overbite | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured vertically from the upper to the lower central incisors' edges (in mm).
Change in the molar relationship | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from the mesial cusp of the maxillary first permanent molar to the mesial cusp of the mandibular first permanent molar (in mm).
Change in the position of the maxillary base | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from A point to a vertical reference plane (in mm).
Change in the position of the mandibular base | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from Pogonion Point to a vertical reference plane (in mm).
Change in the mandibular position relative to the upper jaw | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from A point to Pogonion Point (in mm).
Change in condylar head position | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from Condylion point to the vertical reference plane (in mm).
Change in the composite mandibular length | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from Condylion Point to the Pogonion Point (in mm).
Change in position of the maxillary incisor | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from the upper central incisor edge to the A Point (in mm).
Change in position of the mandibular incisor | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from the lower central incisor edge to the Pogonion Point (in mm).
Change in position of the maxillary permanent first molar | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from the mesial cusp of the maxillary first permanent molar to A Point (in mm).
Change in position of the mandibular permanent first molar | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from the mesial cusp of the mandibular first permanent molar to the Pogonion Point (in mm).
Change in the ramus height | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. The distance was measured vertically from the Articular Point (Ar) to the Gonion Point (Go) in millimeters.
Change in the corpus length | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This was measured sagittally from the Gonion (Go) Point to the Mention (Me) Point. The distance is measured in mm.
Change in MM angle | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This angle, measured in degrees, represented the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis. It is calculated for the internal angle formed by the intersection between the maxillary and mandibular planes.
Change in the SN-OP | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This angle, measured in degrees, represented the relationship between the occlusal plane (OP) and the anterior cranial base (the distance between Sella (S) and Nasion (N)) in the vertical direction.
Change in the SN-MP | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient This angle, measured in degrees, represented the relationship between the lower jaw plane and the cranial base in the vertical direction.
Change in the Bjork sum (N-S-Ar + S-Ar-Go +Ar-Go-Me) | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This angle, measured in degrees, was the sum of three angles: the saddle angle (N-S-Ar angle), the articular angle (S-Ar-Go), and the gonial angle (Ar-Go-Me).
Change in the inclination of the upper incisors. | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This angle, measured in degrees, represented the relationship between the upper incisor axis and the anterior cranial base in the anteroposterior direction. It was measured between the upper incisor axis and the SN plane.
Change in the L1-MP angle | T0: One day before the beginning of the functional treatment, T1: After completing functional treatment which which is expected within 11 months.
  Lateral cephalometric images were taken for each patient. This angle, measured in degrees, represented the relationship between the lower incisor axis and the mandibular base in the anteroposterior direction. It was measured between the lower incisor axis and the Go-Me plane.

CONTACTS AND LOCATIONS:
Overall Officials: Rabea A Ghareeb, DDS, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria; Kinda Sultan, DDS MSc PhD, Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Department of Orthodontics, Faculty of Dentistry, Damascus University
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdulhadi A, Burhan AS, Hajeer MY, Hamadah O, Mahmoud G, Nawaya FR, Namera MO. Evaluation of the Functional Treatment of Patients With Skeletal Class II Malocclusion Using Low-Level Laser Therapy-Assisted Twin-Block Appliance: A Three-Arm Randomized Controlled Trial. Cureus. 2022 Mar 24;14(3):e23449. doi: 10.7759/cureus.23449. eCollection 2022 Mar. PMID 35345811
- [Background] Burhan AS, Nawaya FR. Dentoskeletal effects of the Bite-Jumping Appliance and the Twin-Block Appliance in the treatment of skeletal Class II malocclusion: a randomized controlled trial. Eur J Orthod. 2015 Jun;37(3):330-7. doi: 10.1093/ejo/cju052. Epub 2014 Oct 8. PMID 25296729
- [Background] Tripathi T, Singh N, Rai P, Gupta P. Mini-implant-supported twin-block appliance: An innovative modification. Niger J Clin Pract. 2019 Mar;22(3):432-438. doi: 10.4103/njcp.njcp_342_18. PMID 30837435
- [Background] O'Brien K, Wright J, Conboy F, Sanjie Y, Mandall N, Chadwick S, Connolly I, Cook P, Birnie D, Hammond M, Harradine N, Lewis D, McDade C, Mitchell L, Murray A, O'Neill J, Read M, Robinson S, Roberts-Harry D, Sandler J, Shaw I. Effectiveness of early orthodontic treatment with the Twin-block appliance: a multicenter, randomized, controlled trial. Part 1: Dental and skeletal effects. Am J Orthod Dentofacial Orthop. 2003 Sep;124(3):234-43; quiz 339. doi: 10.1016/S0889540603003524. PMID 12970656
- [Background] Ehsani S, Nebbe B, Normando D, Lagravere MO, Flores-Mir C. Short-term treatment effects produced by the Twin-block appliance: a systematic review and meta-analysis. Eur J Orthod. 2015 Apr;37(2):170-6. doi: 10.1093/ejo/cju030. Epub 2014 Jul 22. PMID 25052373
- [Derived] Ghareeb RA, Sultan K, Hajeer MY, Ajaj MA, Alzoubi H. Comparison of skeletal and dentoalveolar effects of mini-implant-supported twin block versus conventional twin block in treating growing patients with Class II Division 1 malocclusion: a two-arm randomized controlled clinical trial. Eur J Orthod. 2025 Oct 16;47(6):cjaf093. doi: 10.1093/ejo/cjaf093. PMID 41347939